CLINICAL TRIAL: NCT06173505
Title: A Phase 1b/2, Open-label, Randomized Study of Vudalimab in Combination With Chemotherapy or Pembrolizumab in Combination With Chemotherapy as First-line Treatment in Patients With Advanced Non-small Cell Lung Cancer
Brief Title: Study of Vudalimab or Pembrolizumab in Combination With Chemotherapy as First-line Treatment in Patients With Advanced NSCLC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xencor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XmAb717-06
Record Dates: First submitted 2023-11-13; First posted 2023-12-15 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Nonsquamous Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer; Nonsquamous; XmAb20717; vudalimab; anti-PD-1 x anti-CTLA-4; checkpoint inhibitor; chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Pemetrexed; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vudalimab + Carboplatin + Pemetrexed (Experimental)
  Interventions: Combination Product: Vudalimab + Carboplatin + Pemetrexed
- Pembrolizumab + Carboplatin + Pemetrexed (Active Comparator)
  Interventions: Combination Product: Pembrolizumab + Carboplatin + Pemetrexed

INTERVENTIONS:
Combination Product: Vudalimab + Carboplatin + Pemetrexed — Vudalimab intravenous + carboplatin intravenous + pemetrexed intravenous
  Arms: Vudalimab + Carboplatin + Pemetrexed
Combination Product: Pembrolizumab + Carboplatin + Pemetrexed — Pembrolizumab intravenous + carboplatin intravenous + pemetrexed intravenous
  Arms: Pembrolizumab + Carboplatin + Pemetrexed

SUMMARY:
The purpose of this study is to identify the recommended dose of vudalimab to be used in combination with chemotherapy (Part 1) and to evaluate the efficacy and safety of vudalimab plus standard of care chemotherapy relative to pembrolizumab plus chemotherapy (Part 2) as first-line treatment in patients with nonsquamous non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This is a Phase 1b/2 study, multicenter, open-label, randomized study in patients with nonsquamous non-small cell lung cancer without prior treatment for metastatic disease. Part 1 is designed to identify the recommended Phase 2 dose (RP2D) of vudalimab, an anti-PD-1/CTLA-4 bispecific antibody, in combination with standard of care (SOC) chemotherapy. Part 2 will evaluate the efficacy and safety vudalimab, at the RP2D, plus SOC relative to pembrolizumab (anti-PD-1) plus SOC chemotherapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed, locally advanced (unresectable) or metastatic nonsquamous NSCLC
* Documented absence of tumor activating EGFR mutation, ALK gene and ROS1 rearrangements, and alterations in any actionable driver oncogenes for which there are locally approved targeted first-line therapies
* PD-L1 IHC testing documenting TPS < 49%
* No prior systemic treatment for advanced/metastatic NSCLC.
* Measurable disease by RECIST 1.1
* ECOG performance status score of 0 or 1
* Life expectancy ≥ 3 months
* Adequate liver, kidney, thyroid and bone marrow function

Key Exclusion Criteria:

* Have known active central nervous system metastases and/or carcinomatous meningitis. Patients with treated brain metastases may participate, provided they are radiologically stable
* Active known or suspected autoimmune disease
* Has any condition requiring systemic treatment with corticosteroids, prednisone equivalents, or other immunosuppressive medications within 14 days prior to first dose of study drug
* Interstitial lung disease that is symptomatic
* Known human immunodeficiency virus (HIV) positive with CD4+ T-cell (CD4+) count < 350 cells/μL, or an HIV viral load greater than 400 copies/mL, or a history of an acquired immunodeficiency syndrome-defining opportunistic infection within the past 12 months, or not on established antiretroviral therapy (ART) for at least 4 weeks prior to initiation of study drug dosing. (HIV positive subjects who do not meet these exclusion criteria are eligible)
* Positive test for hepatitis C RNA (a patient who is hepatitis C virus [HCV] antibody positive but HCV RNA negative due to documented, curative prior antiviral treatment or natural resolution is eligible)
* Positive test for hepatitis B surface antigen or hepatitis B core antibody (hBcAb) (a patient whose hBsAg is negative and hBcAb is positive may be enrolled if a hepatitis B virus (HBV) DNA test is negative and the subject is retested for HbsAg and HBV DNA every 2 months)
* History or evidence of any clinically unstable/uncontrolled disorder, condition, or disease (including, but not limited to, cardiopulmonary, renal, metabolic, hematologic, or psychiatric) other than NSCLC, that, in the opinion of the Investigator, would pose a risk to patient safety or interfere with study evaluations, procedures, or completion

Other protocol defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Part 1: Recommended Phase 2 dose of vudalimab in combination with chemotherapy | Day 1 to Day 21
  Incidence of treatment-emergent adverse events and treatment-related adverse events leading to discontinuation of treatment
Part 2: Progression free survival | Day 1 to 2.5 years
  Progressive disease per RECIST 1.1 or death, whichever comes first

SECONDARY OUTCOMES:
Antitumor activity | Day 1 to 1.4 years
  Objective response rate as determined by investigator, duration of response (Part 1 and Part 2)
Changes in circulating tumor DNA (ctDNA) | Day 1 to 1.4 years
  Examine ctDNA changes as a surrogate marker for disease burden (Part 1 and Part 2)
Maximum Serum Drug Concentration (Cmax) | Day 1 to 1.4 years
  (Part 1 and Part 2)
Trough Serum Drug Concentration (Ctrough) | Day 1 to 1.4 years
  (Part 1 and Part 2)
Area Under the Concentration-time Curve (AUC) | Day 1 to 1.4 years
  (Part 1 and Part 2)
Overall survival | Day 1 to 2.5 years
  Time to death from any cause (Part 2)
Incidence of treatment-emergent adverse events | Time Frame: Day 1 to 1.4 years]

CONTACTS AND LOCATIONS:
Overall Officials: Jolene Shorr, Study Director — Executive Director, Clinical Development
Locations (43):
- United States (15):
  - Palo Verde Cancer Specialists, Glendale, Arizona
  - Western Regional Medical Center, Goodyear, Arizona
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Mid Florida Hematology and Oncology Center, Orange City, Florida
  - Memorial Cancer Institute at Memorial Hospital West, Pembroke Pines, Florida
  - Midwestern Regional Medical Center, Zion, Illinois
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Minnesota Oncology Hematology, P.A., Maple Grove, Minnesota
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - New Jersey Center for Cancer Research, Brick, New Jersey
  - Cancer Institute at Phelps, Sleepy Hollow, New York
  - Consultants in Medical Oncology and Hematology, P.C., Broomall, Pennsylvania
  - Alliance Cancer Specialists, Horsham, Pennsylvania
  - Hematology Associates of Fredericksburg, Fredericksburg, Virginia
- Jessa Ziekenhuis - Campus Virga Jesse, Hasselt, Belgium
- Greece (2):
  - Athens Medical Center, Athens
  - St. Lukes (Agios Loucas) Hospital, Thessaloniki
- Malaysia (6):
  - Hospital Canselor Tuanku Muhriz, Cheras
  - Pantai Hospital Ipoh, Ipoh
  - Hospital Sultan Ismail, Johor Bahru
  - Hospital Umum Sarawak, Kuching
  - Institut Kanser Negara, Putrajaya
  - Columbia Asia Hospital Bukit Rimau, Shah Alam
- The Netherlands Cancer Institute - Antoni van Leeuwenhoek, Amsterdam, North Holland, Netherlands
- Med-Polonia Sp. Z o.o., Poznan, Poland
- Portugal (3):
  - ULS do Alto Ave, EPE - Hospital da Senhora da Oliveira Guimarães, Guimarães
  - Hospital Santo António dos Capuchos - Unidade Local de Saúde de São José, Lisbon
  - Instituto Português de Oncologia de Porto Francisco Gentil, E.P.E., Porto
- Spain (11):
  - NEXT Oncology-Hospital Quirónsalud Barcelona, Barcelona
  - Hospital Universitario Vall d'Hebrón, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Institut Català d'Oncolgia de Girona, Girona
  - Hospital Clínico San Carlos, Madrid
  - START MADRID-Hospital Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - NEXT Oncology-Hospital Quirónsalud Madrid, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Y Politécnico La Fe, Valencia
- Taiwan (3):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan